CLINICAL TRIAL: NCT07152652
Title: Physiological, Hormonal, and DNA-based Mechanisms of Psychosocial Stress and Therapeutic Effect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Strategic Research Council, Finland (Unknown); University of Eastern Finland (Other); Finnish Institute for Health and Welfare (Other Government); Finnish Cultural Foundation (Other)
Responsible Party: Principal Investigator, Jari Lahti, Professor, University of Helsinki
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 60/2025
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Well-Being, Psychological; Loneliness
Keywords: University Students; Group Intervention; Mental Health; Loneliness; Social Isolation; Anxiety; Depression; Social Anxiety; Social Cohesion; Groups 4 Health; Stress system functioning; Genetics; Epigenetics; Experience Sampling Method; Stress physiology
MeSH Terms: conditions — Psychological Well-Being; Social Isolation; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groups 4 Health Intervention (Experimental): This group will receive the G4H intervention immediately after randomization
  Interventions: Behavioral: Groups 4 health
- Waitlist Control Group (No Intervention): This group will receive the G4H intervention after the 19 weeks waitlist period

INTERVENTIONS:
Behavioral: Groups 4 health — Groups 4 Health (G4H) at the University of Helsinki is a manualized group intervention for the students that focuses on social connectedness and aims at improving general health and life satisfaction. G4H groups are facilitated by two psychology master's students (or licensed psychologists) carefully trained for the intervention and mentored by experienced clinical psychologists. G4H consists of five 90 minutes sessions that aim to give participants the knowledge and skills they need to effectively manage their social group memberships and identities. Each session contains exercises and discussions described in the G4H workbook that target different aspects of group life identified within the social identity model of identity change and put the Social Identity Approach to Health -model to practice. Students earn 2 European Credit Transfer and Accumulation System (ECTS) credits for completing the intervention.
  Other Names: G4H; Ryhmät kuntoon
  Arms: Groups 4 Health Intervention

SUMMARY:
The goal of this trial is to learn if the Groups 4 Health (G4H) intervention is effective in supporting student well-being at the University of Helsinki. It will also learn about the factors that may influence the efficacy of the intervention (such as facilitators characteristics, stress physiology and changes in gene expression). The main questions it aims to answer are:

1. Is the G4H intervention effective and cost-effective in supporting student well-being?
2. To what extent participants' physiological, hormonal, or molecular characteristics mediate the therapeutic effect of the G4H
3. To what extent participants' genotype moderates the effect of the G4H
4. To what extent facilitators' characteristics mediate or moderate the effect of the G4H

Data is collected from both the intervention participants and the facilitators.

The G4H facilitators will:

* Facilitate the G4H intervention.
* Fill in questionnaires and provide physiological and molecular measurements before, during, and after the G4H intervention.

The G4H participants will:

* Participate in the G4H intervention.
* Fill in questionnaires and provide physiological, hormonal and molecular measurements before, during, and after the G4H intervention.

DETAILED DESCRIPTION:
This study is a randomized waitlist-controlled trial for investigating the efficacy and cost-efficacy of Groups 4 Health (G4H) brief psychosocial intervention for loneliness among the students at the University of Helsinki. Furthermore, several biological and psychosocial mechanisms that may exert the effects of psychosocial stress and therapeutic change are studied. In addition to various psychosocial factors, the mechanisms include genetic factors and epigenetic alterations, hypothalamic-pituitary axis (HPA) activity (cortisol), and parasympathetic (heart rate variability) and sympathetic (alpha amylase) function of the autonomic nervous system (ANS).

This trial will investigate:

1. The efficacy and cost-efficacy of the G4H in a wait-list randomized controlled trial (RCT)
2. To what extent participants' physiological, hormonal or molecular measures of ANS, cortisol, alpha amylase, and Deoxyribonucleic Acid methylation (DNAm) mediate the therapeutic effect of the G4H.
3. To what extent participants' genotype moderates the effects of the G4H.
4. To what extent facilitators' characteristics mediates or moderates the effect of the G4H.

The participants will be randomized to start the G4H immediately after randomization or after the waitlist-period of 19 weeks (7 weeks active G4H + 3 months follow-up). The G4H includes five facilitated group sessions and will be delivered over a 7-week period. Data is collected before, during, and after the intervention, as well as in 1-, 3-, and 12-month follow-ups. The waitlist control group does not provide 12-months follow-up data, as they receive the intervention after the 19 weeks waitlist-period.

METHODS:

The study's outcome measures are described in the outcome measures -section. In addition, the following measures are used to answer the research questions.

Experience Sampling Method (ESM):

ESM is used to measure frequent, real-time assessments of participants self-reported mood, and stress appraisals at multiple times throughout the day. ESM is applied to explore the variation and changes in participants daily subjective well-being and loneliness in concurrence with G4H group facilitators stress appraisals before and after facilitation of G4H sessions. The ESM data will be collected using General Data Protection Regulation compliant experience-sampling software program that runs on smartphones (e.g. m-Path).

The daily ESM protocol consists of a morning and evening prompts in which participants are asked to rate their momentarily affect, and daily satisfaction with life. In the morning prompt, participants are also asked to assess daily physiological correlates such as sleep, amount of caffeine, and alcohol consumption, and exercise during the last 24h.

Intervention participants are also asked to answer questions about momentarily appraisal of social company, and loneliness (see outcome measures). Facilitators' event-based sampling takes place before and after the group facilitation and consists of self-report on the appraisals and experiences related to situation with single items derived from widely used questionnaires.

Experiences related to the pre-group situation are assessed from the facilitators during the intervention with items related to momentarily affect: "When thinking about the upcoming group session I feel: calm; happy; determined; enthusiastic; tired; stressed; worried; anxious" (response options: 0 =not at all - 6 = very much), and expectations: "I have prepared well for the session; I trust in my ability to manage the upcoming group session; I expect the session to go well." (response options: 0 = strongly disagree - 6 = strongly agree). Experiences related to the post-group situation are assessed with items related to the group situation: "I feel that the group session went well; I felt competent in facilitating the session; I was present during the session; It was easy for me to feel compassion towards participants" (response options: 0 = strongly disagree - 6 = strongly agree).

Salivary cortisol and alpha amylase:

Saliva samples with Cortisol Salivette synthetic swabs (Sarsted) are collected for cortisol and alpha-amylase measurements from both the intervention participants (see outcomes) and facilitators. These samples are collected by placing a synthetic swab in mouth for 2 minutes and returning it to a plastic tube thereafter.

The cortisol and alpha-amylase samples are provided by the participating facilitators during the first, third, and last intervention sessions. The sampling times are -45, -10, 45, 90, 110, and 135 minutes from the start of the session (6 samples per session).

Covariates related to the stress measurements:

Information on the following potential covariates related to stress physiology is also collected from the intervention participants and facilitators on the same day as the saliva samples are given: situational stress, sleep, physical activity, smoking, alcohol and coffee consumption, menstrual cycle, medication, chronic illness.

Deoxyribonucleic Acid (DNA) measures:

Omnigene saliva Oragene OG-600 DNA (or equivalent) is used for the DNAm and genotype sampling. Both the intervention participants and the facilitators will provide these samples before and immediately after the intervention.

Autonomic nervous system functioning:

A self-developed bra-integrated solution is used to collect non-medical electrocardiogram (ECG)-signal and accelerometer data from the facilitators. Data is collected by wearing a bra during times, when user regularly would use it, but especially on days when there is activity of G4H study. ECG signal is analysed by time- and frequency-based Hearth rate variability analysis (HRV). Accelerometer data is used to estimate physical activity and used for control high movement effects on HRV. HRV is used to assess daily levels of sympathetic and parasympathetic function of the ANS and to estimate cognitive load effects of facilitating G4H sessions.

Participants' background:

Participants' background information is collected from the intervention participants as potential covariates: gender, birth date, mother tongue, marital status, household composition, residential situation, employment status, education, income, subjective financial situation, subjective health, subjective loneliness, subjective minority status and willingness to participate in the intervention and academic skills (4-item organized studying scale, from Learn -questionnaire).

Facilitators' characteristics:

Information is collected at pre-intervention on the facilitator's background (gender, birth date, marital status, household composition, residential situation, employment status, education, work experience, income, subjective financial situation), and professional (12-item Experiences in Close Relationships Short form) and individual (30-item Extra-Short Five -questionnaire) characteristics.

The facilitators will also answer questionnaires during the intervention on study burnout risk (9-item Study Burnout Inventory, at pre-intervention and last session), perceived stress (10-item Perceived Stress Scale, at pre-intervention, 3rd, and last session), self and other compassion (4-item Process Based Assessment Tool, at pre-intervention, 3rd, and last session), and self-assessed skillfulness, difficulties, and feelings (36-item Therapist Work Involvement Scales, at 3rd and last session) as potential mediators or moderators of the intervention's effectiveness.

SAMPLE SIZE AND ANALYSES:

The minimum sample size is 148 intervention participants. Appropriate statistical methods including linear mixed model analyses will be used to study the effectiveness of the G4H intervention and the mediating and moderating factors. Appropriate imputation methods such as multiple imputation by chained equations will be used if necessary.

Written informed consent is gathered from all participants. The participants who have given their consent have the option to withdraw from the study at any point.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and above)
* Student in the University of Helsinki, Finland
* Able to speak/read Finnish, Swedish, or English

Exclusion Criteria:

* None

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Loneliness | 1) Before the intervention, 2) During the intervention (week 3), 3) immediately after the intervention, 4) one month follow-up, 5) three months follow-up, 6) 12 months follow-up
  Loneliness is measured with the 4 and 8-item short forms of the revised University of California, Los Angeles Loneliness Scale (ULS-4 and ULS-8, response options: 1=never, 2=rarely, 3=sometimes, 4=often, lower score means better outcome).
Depression | 1) Before the intervention, 2) immediately after the intervention 3) one month follow-up, 4) three months follow-up, 5) 12-months follow-up
  Symptoms of depression are assessed with the 9-item Patient Health Questionnaire (response options: 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day, lower score means better outcome).
Active group memberships | 1) Before the intervention, 2) During the intervention (week 3), 3) immediately after the intervention, 4) one month follow-up, 5) three months follow-up, 6) 12-months follow-up
  Multiple group memberships are assessed with the 4-item Exeter Identity Transition Scale (response options: 1 = strongly disagree, 7 = strongly agree, higher score means better outcome).
Mental well-being | 1) Before the intervention, 2) immediately after the intervention 3) one month follow-up, 4) three months follow-up, 5) 12-months follow-up
  Mental well-being is assessed with the 7-item Short Warwick-Edinburgh Mental Wellbeing Scale (response options: 1=not at all, 2=rarely, 3=occasionally, 4=often, 5=all the time, higher score means better outcome).
General well-being | 1) Before the intervention, 2) immediately after the intervention 3) one month follow-up, 4) three months follow-up, 5) 12-months follow-up
  General well-being is assessed with the 14-item General Population version of the Clinical Outcomes in Routine Evaluation (response options: 0=not at all, 1=only occasionally, 2=sometimes, 3=often, 4=most of/all of the time, lower score means better outcome).
Anxiety | 1) Before the intervention, 2) immediately after the intervention 3) one month follow-up, 4) three months follow-up, 5) 12-months follow-up
  Symptoms of anxiety are assessed with the 7-item Generalized Anxiety Disorder Questionnaire (response options: 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day, lower score means better outcome).
Social anxiety | 1) Before the intervention, 2) immediately after the intervention 3) one month follow-up, 4) three months follow-up, 5) 12-months follow-up
  Social anxiety is assessed with the 3-item Mini Social Phobia Inventory (response options: 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day, lower score means better outcome).

SECONDARY OUTCOMES:
Perceived Stress | 1) Before the intervention, 2) immediately after the intervention 3) one month follow-up, 4) three months follow-up, 5) 12-months follow-up
  Perceived stress is measured with the 10-item Perceived Stress Scale (response options: 0 = never, 1 = almost never, 2=sometimes, 3=fairly often, 4=very often, lower scores means better outcome)
Self- and other-compassion | 1) Before the intervention, 2) immediately after the intervention 3) one month follow-up, 4) three months follow-up, 5) 12-months follow-up
  Self- and other-compassion is measured with the 4-item Process Based Assessment Tool (response options: 1=very seldom to 5=very often, higher scores means better outcome)
Health-related quality of life | 1) Before the intervention, 2) immediately after the intervention, 3) three months follow-up
  Health-related quality of life is measured with the Euro Quality of Life - 5 dimension - 5 level questionnaire (EQ-5D-5L). The measure has 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) comprising of five statements of which the respondent can choose the option that best describes their situation. Higher score means better outcome. This measure is used to calculate the cost-effectiveness of the interventions.
Use of social and health care services | 1) Before the intervention, 2) immediately after the intervention, 3) three months follow-up
  The use of social and health care services for mental health is measured with a self-report questionnaire (medications, health care appointments, hospitalization, counseling). The use of health care services will be monetarized by using Finnish national unit costs. This measure is used to calculate the cost-effectiveness of the interventions.
Time used by facilitators | Immediately after each intervention session, during 8 weeks
  The time used for planning, executing, and assessing the G4H sessions is reported by the facilitators. This measure is used to calculate the cost-effectiveness of the interventions.
Study credits accumulated over one year | 1 year before the intervention, 1 year after the intervention
  Overall accumulated study credit data is gathered from the University of Helsinki (UH) registries. These data will be used both as measures of effectiveness of the interventions and to account for the confounders in the statistical analyses.
Grade point average | 1 year before the intervention, 1 year after the intervention
  One year grade point average is gathered from the UH registries. These data will be used both as measures of effectiveness of the interventions and to account for the confounders in the statistical analyses.
Weighted grade point average | 1 year before the intervention, 1 year after the intervention
  Weighted grade point average is determined by the grades of each course weighted by the number of credits gained for it.
Study burnout risk | 1) Before the intervention, 2) immediately after the intervention 3) one month follow-up, 4) three months follow-up, 5) 12-months follow-up
  Study burnout risk is measured by the 9-item Study Burnout Inventory (response options: 1=Completely disagree, 2=Disagree, 3=Partly disagree, 4=Partly agree, 5=Agree, 6=Completely agree. Lower score means better outcome).
Sleep quality | 1) Before the intervention, 2) immediately after the intervention 3) one month follow-up, 4) three months follow-up, 5) 12-months follow-up
  Sleep quality is measured with the Single-Item Sleep Quality Scale (response options: 0=terrible to 10=excellent, higher score means better outcome)
Salivary cortisol | The participants provide the samples on two consecutive days 1) before the intervention 2) after the intervention, and 3) at 3-months follow-up. The sampling times are 0, 30, 45, and 60 minutes after awakening (4 samples per day).
  The cortisol awakening profile is used as an index of hypothalamic-pituitary-adrenal axis function reflecting stress physiology. The participants' salivary cortisol profiles are studied relative to awakening times. Atypical awakening profiles indicate poorer outcome.
Salivary alpha-amylase | The participants provide the samples on two consecutive days 1) before the intervention 2) after the intervention, and 3) at 3-months follow-up. The sampling times are 0, 30, 45, and 60 minutes after awakening (4 samples per day). The alpha amylase awake
  The salivary alpha-amylase is used as an index of sympathetic nervous system function reflecting stress physiology. The participants' salivary alpha amylase profiles are studied relative to awakening times. Atypical awakening profiles indicate poorer outcome.
Daily positive and negative affect | 1) Before the intervention, 2) During the intervention, 3) immediately after the intervention, 4) three months follow-up]
  Daily affect is assessed with items of The Positive and Negative Affect Schedule: "To what extent do you currently feel: calm; happy; enthusiastic; tired; stressed; anxious?" (response options: 0 =not at all - 6 = very much).
Daily health-related information | 1) Before the intervention, 2) During the intervention, 3) immediately after the intervention, 4) three months follow-up
  Daily health-related factors are assessed with items adapted from the Finnish Institute of Occupational Health Sleep and Health Information Form. Perceived sleep quality and quantity is assessed with an item "Last night I slept well/ enough". (response options: 0 = strongly disagree - 6 = strongly agree). Use of caffeine, alcohol and nicotine products, and amount of physical activity during the past 24 hours are assessed by reporting usage (yes/ no) or the amounts.
Daily momentary loneliness | 1) Before the intervention, 2) During the intervention, 3) immediately after the intervention, 4) three months follow-up
  Daily momentary loneliness, and appraisals related to company are assessed with items "I feel lonely" (response options: 0 =not at all - 6 = very much), and if in company "I enjoy this company" (response options: 0 = strongly disagree - 6 = strongly agree).
Daily satisfaction with life | 1) Before the intervention, 2) During the intervention, 3) immediately after the intervention, 4) three months follow-up
  Daily life satisfaction is measured with an item: "How satisfied were you with your life today?" (response options: 0 = not at all satisfied - 6 = very satisfied).

OTHER OUTCOMES:
Mood | 1) Before the intervention, 2) During the intervention (week 3), 3) immediately after the intervention, 4) one month follow-up, 5) three months follow-up, 6) 12-months follow-up
  Mood is measured with scale from 0 (extremely bad mood) to 7 (extremely good mood)
Identification with the intervention | During intervention (week 3)
  Identification with the intervention group is assessed with the Single-Item Social Identification -measure (response options: 1 = fully disagree, 7 = fully agree, higher score means better outcome).
Participant adherence | Immediately after each intervention session, during 8 weeks
  The number of participants consented vs the number of participants completing the intervention, attendance rate of individual sessions
Facilitator's fidelity to the manual | Immediately after each intervention session, during 8 weeks
  To monitor fidelity to the G4H manual, the facilitators of the G4H groups will complete a short checklist at the end of each session to determine compliance to the protocol.
Participants' Working alliance | During intervention (week 3)
  Participants' experience of working alliance is assessed with the 12-item Working Alliance Inventory Short and Revised (response options: 1 = never, 2 = rarely, 3 = occasionally, 4 = sometimes, 5 = often, 6 = very often, 7 = always, 3 subscales: goal, task, bond, higher score means better outcome)
Facilitators' Working alliance | During intervention (week 3)
  Facilitators' working alliance is assessed with an 18-item version of the Therapist Working Alliance Inventory Short Form (response options: 1 = never, 2 = rarely, 3 = occasionally, 4 = sometimes, 5 = often, 6 = very often, 7 = always, 3 subscales: goal, task, bond, higher score means better outcome)
Group cohesion | 1) During intervention (week 3), 2) immediately after the intervention
  Group cohesion is measured with the 5-item Group Climate Questionnaire (response options: 0=Not at all, 1=A little bit, 2=Somewhat, 3=Moderately, 4=Quite a bit, 5=A great deal, 6=Extremely, higher score means better outcome).
Completing homework | Immediately after the intervention
  The number of homework assignments completed by the participants is inquired in a questionnaire.
Participants' experiences during the intervention | Immediately after each intervention session, during 8 weeks
  A learning diary is used to collect qualitative description of experiences during the intervention.
Motivation to manage social groups | 1) Before the intervention, 2) during the intervention (week 3), 3) immediately after the intervention
  Motivation to manage social groups is measured by tailored motivation rulers (response options: 1=not at all to 10=extremely, higher score means better outcome)
Treatment motivation | 1) Before the intervention, 2) during the intervention (week 3)
  Treatment motivation is measure by the 16-item Situational Motivation Scale (response options: 1 = corresponds not all, 2 = corresponds very little, 3 = corresponds a little, 4 = corresponds moderately, 5 = corresponds enough, 6 = corresponds a lot, 7 = corresponds exactly, higher score means better outcome)
Social support | 1) Before the intervention, 2) immediately after the intervention
  Social support is measured with the 3 item Social Support Questionnaire (response options Number: 0-9 people giving support, Satisfaction in support: 0 = very dissatisfied, 10 = very satisfied, higher score means better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Helsinki, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haslam C, Cruwys T, Chang MX, Bentley SV, Haslam SA, Dingle GA, Jetten J. GROUPS 4 HEALTH reduces loneliness and social anxiety in adults with psychological distress: Findings from a randomized controlled trial. J Consult Clin Psychol. 2019 Sep;87(9):787-801. doi: 10.1037/ccp0000427. PMID 31403815
- [Background] Haslam C, Cruwys T, Haslam SA, Dingle G, Chang MX. Groups 4 Health: Evidence that a social-identity intervention that builds and strengthens social group membership improves mental health. J Affect Disord. 2016 Apr;194:188-95. doi: 10.1016/j.jad.2016.01.010. Epub 2016 Jan 21. PMID 26828756
- [Background] Haslam C, Holme A, Haslam SA, Iyer A, Jetten J, Williams WH. Maintaining group memberships: social identity continuity predicts well-being after stroke. Neuropsychol Rehabil. 2008 Oct-Dec;18(5-6):671-91. doi: 10.1080/09602010701643449. PMID 18924001
- [Background] Cruwys T, Haslam C, Rathbone JA, Williams E, Haslam SA, Walter ZC. Groups 4 Health versus cognitive-behavioural therapy for depression and loneliness in young people: randomised phase 3 non-inferiority trial with 12-month follow-up. Br J Psychiatry. 2022 Mar;220(3):140-147. doi: 10.1192/bjp.2021.128. PMID 35049477